CLINICAL TRIAL: NCT02856152
Title: A Single-dose, Open-label, Randomized, 4-way Crossover Study to Assess the Relative Bioavailability And Food Effect of a Tablet Formulation of GDC-0276 in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability And Food Effect of a Tablet Formulation of GDC-0276 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The molecule (GDC-276) is no longer in development.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GX29841; 2016-001572-30 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer
MeSH Terms: interventions — GDC-0276

ARMS (4):
- Treatment A Then B Then D Then C (Experimental): Treatment A: a single dose of three 90-mg capsules of GDC-0276 administered orally after at least an 8-hour fast. Treatment B: a single dose of three 90-mg tablets GDC-0276 administered orally after at least an 8-hour fast. Treatment C: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized FDA high-fat meal. Treatment D: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized low-fat meal. Participants will receive Treatment A on Day 1 of first intervention period, followed by Treatment B on Day 1 of second intervention period, followed by Treatment D on Day 1 of third intervention period, and then Treatment C on Day 1 of fourth intervention period. A washout period of 6 days will be maintained between each intervention period.
  Interventions: Drug: GDC-0276 capsule; Drug: GDC-0276 tablets
- Treatment B, Then C, Then A, Then D (Experimental): Treatment A: a single dose of three 90-mg capsules of GDC-0276 administered orally after at least an 8-hour fast. Treatment B: a single dose of three 90-mg tablets GDC-0276 administered orally after at least an 8-hour fast. Treatment C: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized FDA high-fat meal. Treatment D: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized low-fat meal. Participants will receive Treatment B on Day 1 of first intervention period, followed by Treatment C on Day 1 of second intervention period, followed by Treatment A on Day 1 of third intervention period, and then Treatment D on Day 1 of fourth intervention period. A washout period of 6 days will be maintained between each intervention period.
  Interventions: Drug: GDC-0276 capsule; Drug: GDC-0276 tablets
- Treatment C, Then D, Then B, Then A (Experimental): Treatment A: a single dose of three 90-mg capsules of GDC-0276 administered orally after at least an 8-hour fast. Treatment B: a single dose of three 90-mg tablets GDC-0276 administered orally after at least an 8-hour fast. Treatment C: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized FDA high-fat meal. Treatment D: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized low-fat meal. Participants will receive Treatment C on Day 1 of first intervention period, followed by Treatment D on Day 1 of second intervention period, followed by Treatment B on Day 1 of third intervention period, and then Treatment A on Day 1 of fourth intervention period. A washout period of 6 days will be maintained between each intervention period.
  Interventions: Drug: GDC-0276 capsule; Drug: GDC-0276 tablets
- Treatment D, Then A, Then C, Then B (Experimental): Treatment A: a single dose of three 90-mg capsules of GDC-0276 administered orally after at least an 8-hour fast. Treatment B: a single dose of three 90-mg tablets GDC-0276 administered orally after at least an 8-hour fast. Treatment C: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized FDA high-fat meal. Treatment D: a single dose of three 90-mg tablets of GDC-0276 administered orally within 30 minutes of eating a standardized low-fat meal. Participants will receive Treatment D on Day 1 of first intervention period, followed by Treatment A on Day 1 of second intervention period, followed by Treatment C on Day 1 of third intervention period, and then Treatment B on Day 1 of fourth intervention period. A washout period of 6 days will be maintained between each intervention period.
  Interventions: Drug: GDC-0276 capsule; Drug: GDC-0276 tablets

INTERVENTIONS:
Drug: GDC-0276 capsule — Three 90 milligram [mg] capsules of GDC-0276 administered orally.
Drug: GDC-0276 tablets — Three 90 mg GDC-0276 tablets administered orally.

SUMMARY:
This open-label, randomized, 4-way crossover study in healthy participants will determine the relative bioavailability of the tablet formulation relative to the capsule formulation and the effect of a high-fat and low-fat meal on the relative bioavailability of the tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range 18.0 to 32.0 kilograms per meter squared (kg/m^2), inclusive, and a minimum weight of 50.0 kg
* Male participants of reproductive potential must be and willing to continue using medically acceptable contraception and must avoid sperm donation from screening and for at least 90 days after the last study drug administration

Exclusion Criteria:

* Self-reported substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, and/or participants who have ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence
* Have used any prescription or over-the-counter (OTC) medication or supplement within 14 days or 5 times the elimination half-life (whichever is longer) before Day -1 until the end of their participation in the study
* Have used any vaccine within 7 days before GDC-0276 administration
* Female participants with a positive serum or urine pregnancy test or are breast feeding
* Donation or loss of more than 500 milliliter (mL) whole blood within 3 months preceding entry into the treatment period
* Blood transfusion within 30 days preceding entry into the treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Cmax of M12 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Maximum Plasma Concentration (Cmax) of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Cmax of M16 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastu) of M12 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastu) of M16 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] of M12 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Relative Bioavailability: Geometric Mean Ratio (Tablet/Capsule) of Log Transformed Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] of M16 Metabolite of GDC-0276 | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of M12 Metabolite of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of M16 Metabolite of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Apparent Oral Clearance (CL/F) of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Apparent Oral Clearance (CL/F) of M12 Metabolite of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Apparent Oral Clearance (CL/F) of M16 Metabolite of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Apparent Volume of Distribution (Vz/F) of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Apparent Volume of Distribution (Vz/F) of M12 Metabolite of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Plasma Terminal Half-Life (t1/2) of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Plasma Terminal Half-Life (t1/2) of M12 Metabolite of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Plasma Terminal Half-Life (t1/2) of M16 Metabolite of GDC-0276 Following High-fat Meals, low-fat Meals and in Fasted State on a Tablet Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose
Number of Participants With Adverse Events and Serious Adverse Event | Baseline up to Follow up (Day 32)
Apparent Volume of Distribution (Vz/F) of M16 Metabolite of GDC-0276 Following Tablet and Capsule Dosing | Pre-dose (within 0.5 hours of dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144 hours post-Day 1, or Day 7, or Day 13, or Day 19 dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom